CLINICAL TRIAL: NCT00000704
Title: A Multicenter Dose Ranging Clinical Trial of 2',3'-Dideoxycytidine in the Treatment of Patients With AIDS and Advanced ARC.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 012; 10988 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Antigens; Immunologic Surveillance; Zalcitabine; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; CD4-Positive T-Lymphocytes
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zalcitabine

INTERVENTIONS:
Drug: Zalcitabine

SUMMARY:
To evaluate the long-term safety and effectiveness of the drug 2',3'-dideoxycytidine ( zalcitabine; ddC ) in treating patients with AIDS or advanced AIDS related complex ( ARC ).

Recent studies show that a certain group of drugs (dideoxynucleosides) are effective in treating patients with HIV infection. ddC is a dideoxynucleoside and test tube studies show that it may be valuable in treating AIDS patients. ddC has been shown to be well tolerated in certain patients with AIDS.

DETAILED DESCRIPTION:
Recent studies show that a certain group of drugs (dideoxynucleosides) are effective in treating patients with HIV infection. ddC is a dideoxynucleoside and test tube studies show that it may be valuable in treating AIDS patients. ddC has been shown to be well tolerated in certain patients with AIDS.

A range of doses of ddC is given to patients with AIDS and ARC. Eight patients with AIDS and eight patients with ARC are given ddC at the lowest level for 12 weeks. Patients who respond with a rise in their number of T4 cells or with a fall in HIV antigen in their serum (the fluid portion of the blood) are continued at that dose for an additional 12 weeks. Patients who do not respond at a given dose level (no rise in T4 or fall in serum HIV antigen) stop treatment at 12 weeks. All patients are followed off therapy for 4 weeks. As each dose level is found to be well tolerated for 10 weeks in five of the eight patients in each group, additional patients will be entered at higher dose levels until eight AIDS and eight ARC patients are receiving the drug at a given level.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aspirin, acetaminophen, and nonsteroidal anti-inflammatory agents.
* Acute therapy (7 days) with oral acyclovir.
* Acute therapy with ketoconazole.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Negative antigen test within 2 weeks of starting therapy.
* Significant malabsorption (> 10 percent weight loss within past 3 months with serum carotene < 75 IU/ml or vitamin A < 75 IU/ml).
* Significant cardiac, liver, or neurologic disease.
* For group A:
* Opportunistic infection or malignancy fulfilling definition of AIDS, or with concurrent neoplasm other than basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* For group B:
* Active opportunistic infection, symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to study entry, or with concurrent neoplasms other than KS, basal cell carcinoma of the skin, or in situ carcinoma of the cervix.

Concurrent Medication:

Excluded:

* Acyclovir therapy.
* Chemoprophylaxis for Pneumocystis carinii pneumonia.
* Other antiretroviral agents, biologic modifiers, or systemic corticosteroids.
* Other experimental medications, sedatives, and barbiturates.
* Group B:
* Therapy and/or prophylaxis for AIDS-defining opportunistic infection, antineoplastic therapy.

Concurrent Treatment:

Excluded:

- Transfusion dependency (requiring 2 units of blood more than once per month). Patients with history of idiopathic thrombocytopenia purpura are excluded.

Prior Medication:

Excluded within 30 days of study entry:

* Biologic modifiers or corticosteroids.
* Excluded within 90 days of study entry:
* Antiretroviral agents.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Transfusion.

Inclusion criteria are:

* Consistently positive HIV antigen as defined by Abbott HIV antigen test. This demonstration will be seen on two occasions, each separated by at least 72 hours, the last of which must be within 2 weeks of starting therapy.
* HIV antigen titer must be = or > 100 pg.
* Positive antibody to HIV confirmed by any federally licensed enzyme-linked immunosorbent assay (ELISA) test kit.

The following conditions are allowed:

- Basal cell carcinoma of the skin or in situ carcinoma of the cervix. Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Study Completion 1990-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merigan TC, Study Chair
Locations (1):
- Univ. of Miami AIDS CRS, Miami, Florida, United States

REFERENCES:
- [Background] Merigan TC, Skowron G, Bozzette SA, Richman D, Uttamchandani R, Fischl M, Schooley R, Hirsch M, Soo W, Pettinelli C, et al. Circulating p24 antigen levels and responses to dideoxycytidine in human immunodeficiency virus (HIV) infections. A phase I and II study. Ann Intern Med. 1989 Feb 1;110(3):189-94. doi: 10.7326/0003-4819-110-3-189. PMID 2536257
- [Background] Merigan TC, Skowron G. Safety and tolerance of dideoxycytidine as a single agent. Results of early-phase studies in patients with acquired immunodeficiency syndrome (AIDS) or advanced AIDS-related complex. Study Group of the AIDS Clinical Trials Group of the National Institute of Allergy and Infectious Diseases. Am J Med. 1990 May 21;88(5B):11S-15S. doi: 10.1016/0002-9343(90)90415-a. PMID 2159703